CLINICAL TRIAL: NCT00102999
Title: Impaired Motor Learning and LTP/LTD-like Plasticity in Dystonia, Are Associated With Abnormal Modulation of Cortical Excitability by Somatosensory Volleys
Brief Title: Brain Function in Focal Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050094; 05-N-0094
Record Dates: First submitted 2005-02-04; First posted 2005-02-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-01-22

CONDITIONS: Dystonia
Keywords: Learning; PAS; Upper Limb; TMS; Somatosensory; Dystonia; Upper Limb Dystonia; Healthy Volunteer; HV
MeSH Terms: conditions — Dystonia

SUMMARY:
Objectives

The main objectives of this proposal are (1) to characterize motor learning abnormalities in patients with focal dystonia; (2) to show, using transcranial magnetic stimulation, that this abnormal motor learning went together with an impaired modulation by somatosensory inputs of short and long-interval paired-pulse inhibitions (sICI, lICI) and facilitations (sICF, ICF) of MEPs (ICIs and ICFs are thought to reflect activity of inhibitory and excitatory interneuron's in the primary motor cortex M1); (3) to show that abnormalities of long-term potentiation and long-term depression (LTP/LTD)-like mechanisms (tested using a paired associative stimulation (PAS) intervention), thought to play a crucial role in learning, are associated in dystonia with an abnormal modulation of ICIs and ICFs by somatosensory inputs.

Study population

30 patients with a focal upper limb dystonia and 45 healthy volunteers will take part in the main study. 7 patients with a focal upper limb dystonia and 12 healthy volunteers will take part in the control study.

Design

In the main study: subjects will complete 5 different sessions: visit 1: clinical screening, 1 hour; visit PAS session, 3 hours; visit 3: a minimum of 7 days later, motor learning session, 3 hours; visit 4: follow-up 24 hours later, 1 hour and a half; visit 5, follow-up 48 hours later, 1 hour and a half. During the PAS session they will receive 15 minutes of repeated paired stimulations (transcranial magnetic stimulation -TMS- and peripheral stimulation) thought to produce LTP/LTD like phenomena in M1. During the motor learning sessions they will be asked to perform, as fast as possible, a metronome-paced (0.5 Hz) pinch of their index finger and thumb. They will have 3 blocks of motor practice during the motor learning session.

Between each block of motor practice and before and after PAS, while they rest, subjects will receive paired-pulse transcranial magnetic stimulations (TMS) associated or not with peripheral nerve stimulation in order to assess interactions at M1 cortical level between somatosensory incoming volleys and intracortical inhibitory and excitatory interneuron's.

In the control study: subjects will complete a unique session. They will receive a PAS intervention. Before and after the PAS intervention, spinal excitability will be tested by the means of H reflexes evoked in wrist flexor muscles.

Outcome measures:

The behavioral effect of the motor training or of the PAS intervention will be assessed by measuring the mean peak acceleration (MPA) of thumb movement during the blocks of motor practice and the mean maximal peak force (MPF) between the index finger and thumb before and after the blocks of motor practice.

The activity of different sets of intracortical interneurons (short and long interval GABA related inhibitions: sICI, lICI, intracortical glutamate-related facilitation: ICF and short interval facilitation: sICF) can be tested using paired-pulse TMS paradigms. The effect of learning (or of PAS intervention) on the interaction between somatosensory afferent input and intracortical processes will be assessed by comparing the amount of sICI, lICI, ICF and sICF when associated or not with a peripheral nerve stimulation (median and ulnar nerve stimulation) in a trained muscle (flexor pollicis brevis: FPB) and a non-trained muscle (abductor digiti minimi: ADM) at different times during and after the motor learning or the PAS intervention.

The effect of PAS on spinal cord excitability will be assessed by comparing the size of the H reflex before and after PAS.

DETAILED DESCRIPTION:
OBJECTIVES:

The main objectives of this proposal are (1) to characterize motor learning abnormalities in patients with focal dystonia; (2) to show, using transcranial magnetic stimulation, that this abnormal motor learning went together with an impaired modulation by somatosensory inputs of short and long-interval paired-pulse inhibitions (sICI, lICI) and facilitations (sICF, ICF) of MEPs (ICIs and ICFs are thought to reflect activity of inhibitory and excitatory interneurons in the primary motor cortex M1); (3) to show that abnormalities of long-term potentiation and long-term depression (LTP/LTD)-like mechanisms (tested using a paired associative stimulation (PAS) intervention), thought to play a crucial role in learning, are associated in dystonia with an abnormal modulation of ICIs and ICFs by somatosensory inputs.

STUDY POPULATION:

30 patients with a focal upper limb dystonia and 45 healthy volunteers will take part in the main study.

19 patients with a focal upper limb dystonia and 24 healthy volunteers will take part in the control study.

DESIGN:

In the main study: subjects will complete 5 different sessions: visit 1: clinical screening, 1 hour; visit 2: PAS session, 3 hours; visit 3: a minimum of 7 days later, motor learning session, 3 hours; visit 4: follow-up 24 hours later, 1hour and half; visit 5, follow-up 48 hours later, 1 hour and half. During the PAS session they will receive 15 minutes of repeated paired stimulations (transcranial magnetic stimulation -TMS- and peripheral stimulation) thought to produce LTP/LTD like phenomena in M1. During the motor learning sessions, they will be asked to perform, as fast as possible, a metronome-paced (0.5 Hz) pinch of their index finger and thumb. They will have 3 blocks of motor practice during the motor learning session.

Between each block of motor practice and before and after PAS, while they rest, subjects will receive paired-pulse transcranial magnetic stimulations (TMS) associated or not with peripheral nerve stimulation in order to assess interactions at M1 cortical level between somatosensory incoming volleys and intracortical inhibitory and excitatory interneurons.

In the control studies: subjects will complete a maximum of eight sessions. They will receive a PAS intervention. Before and after the PAS intervention, spinal excitability will be tested by the means of H reflexes evoked in wrist flexors muscles; H reflexes will be delivered alone or will be conditioned by cubital or radial nerve stimulation.

OUTCOME MEASURES:

The behavioral effect of the motor training or of the PAS intervention will be assessed by measuring the mean peak acceleration (MPA) of thumb movement during the blocks of motor practice and the mean maximal peak force (MPF) between the index finger and thumb before and after the blocks of motor practice.

The activity of different sets of intracortical interneurons (short and long interval GABA related inhibitions: sICI, lICI, intracortical glutamate-related facilitation: ICF and short interval facilitation: sICF) can be tested using paired-pulse TMS paradigms. The effect of learning (or of PAS intervention) on the interaction between somatosensory afferent input and intracortical processes will be assessed by comparing the amount of sICI, lICI, ICF and sICF when associated or not with a peripheral nerve stimulation (median and ulnar nerve stimulation) in a trained muscle (flexor pollicis brevis: FPB) and a non-trained muscle (abductor digiti minimi: ADM) at different times during and after the motor learning or the PAS intervention.

The effect of PAS on spinal cord excitability will be assessed by comparing the size of the H reflex alone, the amounts of postactivation depression and those of presynaptic inhibition before and after PAS.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy volunteers (aged 18 or older) who are willing to participate.
* Patients (aged 18 and older) with an idiopathic upper limb dystonia, who are able to practice the motor learning task.

EXCLUSION CRITERIA:

* Subjects with a history of neurological or psychiatric disorder, current use or a history of alcohol or drug abuse, psychiatric disorders requiring hospitalization or prolonged treatment such as substance abuser addiction, head injury with loss of consciousness, epilepsy.
* Subjects with significant hearing loss.
* Subjects receiving drugs acting primarily on the central nervous system.
* Subjects who have been treated with botulinum toxin injections 3 months prior to their participation in the study.
* Subjects who are taking any medication for dystonia at the time of the study.
* Subjects who have already participated in a protocol using a motor learning task.
* Subjects who practice intensively playing any kind of music instrument.

The following exclusion criteria are due to the use of transcranial magnetic stimulation:

* Subjects with cardiac pacemakers, intracardiac lines, implanted medication pumps.
* Subjects with eye, blood vessel, cochlear, or eye implants.
* Subjects with increased intracranial pressure as evaluated by clinical means.
* Subjects with metal in the cranium.
* Subjects with dental braces (but dental fillings are not a problem), metal fragments from occupational exposure or surgical clips in or near the brain.

Women in the last trimester of pregnancy will not be studied because they will likely be uncomfortable maintaining a motionless seated posture during the three hour experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118
Dates: Start 2005-01-31; Study Completion 2009-01-22

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Burke RE, Fahn S, Marsden CD, Bressman SB, Moskowitz C, Friedman J. Validity and reliability of a rating scale for the primary torsion dystonias. Neurology. 1985 Jan;35(1):73-7. doi: 10.1212/wnl.35.1.73. PMID 3966004
- [Background] Abbruzzese G, Marchese R, Buccolieri A, Gasparetto B, Trompetto C. Abnormalities of sensorimotor integration in focal dystonia: a transcranial magnetic stimulation study. Brain. 2001 Mar;124(Pt 3):537-45. doi: 10.1093/brain/124.3.537. PMID 11222454
- [Background] Bara-Jimenez W, Catalan MJ, Hallett M, Gerloff C. Abnormal somatosensory homunculus in dystonia of the hand. Ann Neurol. 1998 Nov;44(5):828-31. doi: 10.1002/ana.410440520. PMID 9818942